CLINICAL TRIAL: NCT01154660
Title: Effects of Increased Tidal Volume on Internal Jugular Vein Cross-sectional Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hye-Keum Kil / Professor, Department of Anaesthesiology and Pain Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4-2009-0734
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: General Anesthesia; Surgery
Keywords: any operation that required for general anesthesia
MeSH Terms: interventions — Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neutral (Experimental)
  Interventions: Other: Tidal Volume
- Trendelenberg (Active Comparator)
  Interventions: Other: Tidal Volume

INTERVENTIONS:
Other: Tidal Volume — observation of IJV circumference and cross sectional area using ultrasonography by changing of tidal volume

SUMMARY:
As increasing tidal volume, the cross sectional area and circumference of Internal Jugular Vein (IJV) could increase. And In the previous study, Trendelenburg position can increase size of IJV. So investigators would compare the cross sectional area, circumference of IJV and peak airway pressure in neutral and Trendelenburg position

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing general anesthesia

Exclusion Criteria:

* history of IJV cannulation
* uncontrolled cardiovascular disease
* severe pulmonary problem
* cervical spinal impairment

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Anesthesiology & Pain Medicine, Seoul, South Korea